CLINICAL TRIAL: NCT05503732
Title: Effects of Energy Drinks on Sleep and Cardiovascular Health in Healthy Young Adults A Double Blind Randomized Clinical Trial
Brief Title: Effects of Energy Drinks on Sleep and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anna Svatikova, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 21-012902
Record Dates: First submitted 2022-07-14; First posted 2022-08-17 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Caffeine
Keywords: Energy Drink
MeSH Terms: interventions — Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy drink first, then placebo drink (Experimental): Subjects will consume two 16-oz energy drinks before sleep for the first study visit, then consume two 16-oz identical looking placebo drink before sleep at the second study visit.
  Interventions: Other: Energy Drink; Other: Placebo Drink
- Placebo drink first, than energy drink (Experimental): Subjects will consume two 16-oz identical looking placebo drink before sleep at the fist study visit, then consume two 16-oz energy drinks before sleep for the second study visit.
  Interventions: Other: Energy Drink; Other: Placebo Drink

INTERVENTIONS:
Other: Energy Drink — Two 16-oz energy drinks consumed orally to be finished approximately 4 hours prior to bed
Other: Placebo Drink — Two 16-oz identical looking placebo drink without caffeine consumed orally to be finished approximately 4 hours prior to bed

SUMMARY:
The purpose of this study is to learn about the change in quality of sleep, structural organization of sleep, and cardiovascular responses after consuming an energy drink compared to a placebo drink with no caffeine or stimulants.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older.
* Healthy subjects without known cardiovascular disease and thyroid disease.
* Subjects who are on no medications (except oral contraceptive pill).
* Nonsmokers.
* No prior history of caffeine sensitivity or allergy.

Exclusion Criteria:

* Subjects with known cardiovascular or thyroid disease.
* Subjects currently taking medications other than oral contraceptive pill.
* Smokers.
* Prior history of caffeine sensitivity or allergy.
* Pregnancy.
* Subjects who regularly consume energy drinks.
* Subjects who typically go to sleep after midnight.
* Subjects who traveled across 2 time zones in the last 7 days.
* Shift workers.
* Subjects who have or are suspected to have sleep apnea.
* Subjects who have a body mass index > 35kg/m^2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Changes in sleep efficiency | Throughout duration of sleep on both nights (night 1 and night 2)
  Time asleep / time in bed
Changes in sleep continuity | Throughout duration of sleep on both nights (night 1 and night 2)
  Frequency of wakefulness after sleep initiation
Changes in sleep architecture | Throughout duration of sleep on both nights (night 1 and night 2)
  Time spent in each stage of sleep
QT segment | Baseline, approximately 1 hour prior to energy drink consumption
  QT duration
QT segment | Throughout duration of sleep on both nights (night 1 and night 2)
  QT duration
Atrial arrhythmias | Baseline, approximately 1 hour prior to energy drink consumption
  Frequency of ectopic atrial beats
Atrial arrhythmias | Throughout duration of sleep on both nights (night 1 and night 2)
  Frequency of ectopic atrial beats
Ventricular arrhythmias | Baseline, approximately 1 hour prior to energy drink consumption
  Frequency of ectopic ventricular beats
Ventricular arrhythmias | Throughout duration of sleep on both nights (night 1 and night 2)
  Frequency of ectopic ventricular beats

SECONDARY OUTCOMES:
Sympathetic activation quantified by changes in plasma norepinephrine | Baseline and AM of day 2
  Plasma norepinephrine while supine
Sympathetic activation quantified by changes in plasma epinephrine | Baseline and AM of day 2
  Plasma epinephrine while supine
Sympathetic activation quantified by changes in plasma dopamine | Baseline and AM of day 2
  Plasma dopamine while supine
Sympathetic activation quantified by urine norepinephrine | Approximately 24 hours
  Total urine norepinephrine secretion
Sympathetic activation quantified by urine epinephrine | Approximately 24 hours
  Total urine epinephrine secretion
Sympathetic activation quantified by urine dopamine | Approximately 24 hours
  Total urine dopamine secretion

OTHER OUTCOMES:
Changes in resting heart rate | Baseline and AM of day 2
  Seated heart rate
Changes in resting blood pressure | Baseline and AM of day 2
  Seated systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Anna Svatikova, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States